CLINICAL TRIAL: NCT04137211
Title: Acute Effects of Sitting and Physical Activity on Cerebrovascular Circulation Among Adults
Brief Title: Acute Effects of Sitting and Physical Activity on Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Swedish School of Sport and Health Sciences (Other)
Collaborators: The Knowledge Foundation (Unknown); ICA-gruppen (Unknown); Intrum AB (Unknown); SATS (Unknown); Monark Exercise (Unknown); Itrim (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Dnr:2019-00998
Record Dates: First submitted 2019-10-15; First posted 2019-10-23 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Healthy Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prolonged sitting with social break (Experimental)
  Interventions: Behavioral: Prolonged sitting with social break
- Prolonged sitting with walk break (Experimental)
  Interventions: Behavioral: Prolonged sitting with walk break
- Prolonged sitting with simple resistance activities (Experimental)
  Interventions: Behavioral: Prolonged sitting with simple resistance activities

INTERVENTIONS:
Behavioral: Prolonged sitting with social break — Participants are required to sit for three hours (reading is permitted), with a toilet break in between. Every thirty minutes participants will have a short social break. Test day begins at 7:30 with pretest measures, followed by the intervention at about 9:00, which will end around 12:00, with subsequent posttest measures.
  Arms: Prolonged sitting with social break
Behavioral: Prolonged sitting with walk break — Participants are required to sit for three hours (reading is permitted), with a toilet break in between. Every thirty minutes participants will have a physical activity break, where they will perform a brisk walk for about three minutes on a treadmill at a predetermined speed and grade based on the fitness test performed during the familiarization session. Test day begins at 7:30 with pretest measures, followed by the intervention at about 9:00, which will end around 12:00, with subsequent posttest measures.
  Arms: Prolonged sitting with walk break
Behavioral: Prolonged sitting with simple resistance activities — Participants are required to sit for three hours (reading is permitted), with a toilet break in between. Every thirty minutes participants will have a physical activity break, where they will perform simple resistance activities following a video for about three minutes. Test day begins at 7:30 with pretest measures, followed by the intervention at about 9:00, which will end around 12:00, with subsequent posttest measures.
  Arms: Prolonged sitting with simple resistance activities

SUMMARY:
The specific aim of this study is to understand how a working day composed of prolonged sitting, sitting regularly interrupted by light aerobic exercise or resistance exercise affects an important mechanism underpinning healthy brain functions, namely cerebral blood flow. It is primarily focused on investigating these effects in ecologically valid conditions, i.e. activity patterns that closely resemble a typical day at the office.

DETAILED DESCRIPTION:
The study will be a controlled crossover experimental trial with three conditions involving 13 adult participants aged between 40 and 60 years. Each participant will complete each of the three experimental conditions, separated by a washout period of minimum four days. As well, physical activity behaviours and sleep the day/night before the test day will be measured. The first visit will be a familiarization session. On the second, third, and fourth visits, participants will undergo three different standardized 3-hour interventions in a randomized order. Before and immediately after the three-hour interventions, blood pressure, augmentation index, and cerebral hemodynamic response of the prefrontal cortex during standardized cognitive tasks (1,2, and 3-back tests) will be measured. Additionally, saliva samples will be collected the morning of the test day and before and after the interventions, blood glucose will be assessed continuously during the trial, and fitness will be measured at the familiarization visit.

ELIGIBILITY:
Inclusion Criteria:

- Has a BMI under 35kg/m2

Exclusion Criteria:

* Has diabetes, epilepsy, or circulatory conditions
* Has experienced heart failure, stroke, or myocardial infarction
* Takes treatment for high blood pressure, sleep disorders, depression, or psychosis

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Changes in cerebral blood flow | before to after 3 hour intervention
  Oxygenated and deoxygenated hemoglobin concentration changes measured with functional near-infrared spectroscopy

SECONDARY OUTCOMES:
Augmentation index | before to after 3 hour intervention
  as a measure of arterial stiffness
Blood glucose levels | during the 3 hour intervention
Cortisol | before to after 3 hour intervention
Mood | before to after 3 hour intervention
  measured with the Positive and Negative Affect Schedule (PANAS) comprised of 20 affect states (10 positive and 10 negative), each affect state scored on a scale going from 1 (very slightly or not at all) to 5 (extremely)
Sleepiness | before to after 3 hour intervention
  measured with Karolinska Sleepiness Questionnaire; goes from 1 (extremely alert) to 9 (extremely sleepy)
Cognitive performance | before to after 3 hour intervention
  nback cognitive test (time and accuracy)
Alertness | before to after 3 hour intervention
  measured with a Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ekblom, PhD, Principal Investigator — The Swedish School of Sport and Health Sciences (GIH)
Locations (1):
- The Swedish School of Sport and Health Sciences (GIH), Stockholm, Sweden

REFERENCES:
- [Derived] Heiland EG, Tarassova O, Fernstrom M, English C, Ekblom O, Ekblom MM. Frequent, Short Physical Activity Breaks Reduce Prefrontal Cortex Activation but Preserve Working Memory in Middle-Aged Adults: ABBaH Study. Front Hum Neurosci. 2021 Sep 16;15:719509. doi: 10.3389/fnhum.2021.719509. eCollection 2021. PMID 34602995